CLINICAL TRIAL: NCT01397773
Title: The Role Pentraxin-3 in the Inflammatory Process in Chronic Renal Failure, and the Association With Other Inflammatory Parameters
Brief Title: Pentraxin-3 in Chronic Renal Failure
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Meltem Gursu, Haseki Training and Research Hospital
Other Study IDs: PTX-HASEKI
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Inflammation; Chronic Kidney Disease
Keywords: Hemodialysis; peritoneal dialysis; chronic kidney disease; inflammation; carotis intima media thickness
MeSH Terms: conditions — Inflammation; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hemodialysis group: Patients on chronic hemodialysis program
- Peritoneal dialysis group: Patients on chronic peritoneal dialysis program
- Pre-dialysis group: Patients with chronic kidney disease stage-4
- Control group: Healthy subjects

SUMMARY:
The aim of the study is to measure Pentraxin-3 levels in patients on hemodialysis, peritoneal dialysis and those in the pre-dialysis period; and to compare these groups with the control group; so as to investigate the eligibility of it as a reliable marker of inflammation; relationship with other inflammatory markers and carotis intima media thickness.

DETAILED DESCRIPTION:
The investigators planned to involve four group of patients: Hemodialysis, peritoneal dialysis, pre-dialysis and the control group; with about 25 patients planned to be involved in each group. The laboratory parameters to be measured are Pentraxin-3, C-reactive protein (CRP), high sensitive CRP, fibrinogen and interleukin-6. Concomitantly, carotis intima media thickness will be measured in the radiology clinic. Statistical analysis will be carried on by Statistical Package for Social Sciences (SPSS) for Windows 13.0. The variables acting on the inflammatory parameters and the correlation between them and carotis intima media thickness will be studied.

ELIGIBILITY:
Inclusion Criteria:

* To give informed consent
* Hemodialysis or peritoneal dialysis for more than 3 months
* Creatinin clearance less than 30 ml/min for the pre-dialysis group

Exclusion Criteria:

* Not to give informed concent
* Active infection within the last 3 months
* Known chronic inflammatory disease

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected among those who are followed up in our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pentraxin-3 level | Five months
  Pentraxin-3 level will be compared with other inflammatory markers.

SECONDARY OUTCOMES:
Carotis intima media thickness | Five months
  Correlation of Pentraxin-3 and carotis intima media thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)